CLINICAL TRIAL: NCT05109793
Title: Prospective Longitudinal Study of Neurological Disease Trajectory in Children Living With Late-Infantile or Juvenile Onset of GM1 or GM2 Gangliosidosis
Brief Title: GM1 and GM2 Gangliosidosis PROspective Neurological Disease TrajectOry Study (PRONTO)
Acronym: PRONTO
Status: Completed | Type: Observational
Sponsor: Azafaros A.G. (Industry)
Responsible Party: Sponsor
Other Study IDs: AZA-001-5A4-01
Record Dates: First submitted 2021-10-08; First posted 2021-11-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: GM1 Gangliosidosis; Sandhoff Disease; Tay-Sachs Disease
Keywords: GM1 Gangliosidosis; GM2 Gangliosidosis; Natural History Study; Lysosomal Storage Disorders; Nervous System Diseases; Tay-Sachs disease; Sandhoff disease; Genetic Diseases, Inborn; Hexosaminidase A and B deficiency; β-galactosidase deficiency
MeSH Terms: conditions — Gangliosidosis, GM1; Sandhoff Disease; Tay-Sachs Disease; Gangliosidoses, GM2; Lysosomal Storage Diseases; Nervous System Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Late infantile or juvenile onset for GM1 or GM2 Gangliosidosis. The study anticipates to include a total of approximately 35 patients.

SUMMARY:
The study aims to characterize prospectively longitudinal progression of neurological domains in GM1 and GM2 Gangliosidosis patients with high-quality standards (GCP compliant).

DETAILED DESCRIPTION:
The study is a prospective longitudinal, multicentric decentralized trial which will be performed in children diagnosed with late infantile or juvenile onset of neurological disease of either GM1 or GM2 Gangliosidoses (Tay-Sachs or Sandhoff disease). The study anticipates to include a total of approximately 35 patients. A large set of neurological functions will be evaluated by rating scales used by physicians and questionnaires answered by parents. Digital tools will be used to support the study procedures with virtual visits.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed GM1 Gangliosidosis or genetically confirmed Tay-Sachs or Sandhoff disease
* Onset of neurological symptoms on or after the patient's first birthday
* Achieved 12-month developmental milestones at normal developmental time points as per Principal Investigator's judgement
* Abnormal gait and/or speech disturbance

Exclusion Criteria:

* Patients who have received (within 6 months before screening), are currently receiving or are planned to receive (within the following 6 months) gene therapy, stem cell transplantation, experimental drugs, or any drug, which, in the Investigator´s opinion, may (have) interfere(d) with disease progression

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with diagnosis of GM1 Gangliosidosis Tay-Sachs disease, or Sandhoff disease, or late infantile or juvenile onset of neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Change in the Gait 9-point item score of the Scale for Assessment and Rating of Ataxia (SARA) | 0-4 years
  Score between 0 (better) and 8 (worse) points
Change in the Speech 7-point item score of SARA | 0-4 years
  Score between 0 (better) and 6 (worse) points

OTHER OUTCOMES:
Change in scores of SARA items Stance (7-point), Sitting (5-point), Finger chase (5-point), Nose-finger test (5-point), Fast alternating hand movement (5-point), Heel-shin slide (5-point) and overall score. | 0-4 years
  Stance score between 0 (better) and 6 (worse) points Sitting score between 0 (better) and 4 (worse) points Finger chase test score between 0 (better) and 4 (worse) points Nose-finger test score between 0 (better) and 4 (worse) points Fast alternating hand movements test score between 0 (better) and 4 (worse) points Heel-shin slide score between 0 (better) and 4 (worse) points
Change in the total score of the Motor Function Measure-32 (MFM-32), and each of the 3 domains | 0-4 years
  The scoring of each item uses a 4-point Likert scale - score between 0 (worse) and 3 (better)
Change of Timed Up & Go | 0-4 years
  Time a patient takes to rise from a chair, walk 3 meters, turn around 180°, walk back to the chair, and sit down while turning 180°
Change in swallowing score | 0-4 years
  Assessment of patient swallowing ability - score between 0 (better) and 5 (worse)
Change in the overall composite score of the Vineland Adaptive Behavioral Scale (VABS) | 0-4 years
  Rated on 0 (never performed),1, 2 (habitually performed) scale
Change in BSFC-s score for each of the 10 items and overall score | 0-4 years
  Rated on a 4-point scale with the values "strongly disagree", "disagree", "agree", and "strongly agree"
Collection of seizures events, choking episodes, respiratory tract infections | 0-4 years
  Gathering data about presence/absence and frequency of seizures, choking episodes, respiratory tract infections

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Mayo Clinic Rochester, Rochester, Minnesota
- Brazil (2):
  - Hospital Pequeno Principe, Curitiba
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
- France (3):
  - Hopital d'Enfants CHU Timone, Marseille
  - Armand-Trousseau Children's Hospital - CHU Paris Est, Paris
  - Hôpital des Enfants - CHU Toulouse Purpan, Toulouse
- Germany (2):
  - Universtitäsklinikum Giessen und Marburg, Giessen
  - LMU - Klinikum der Universitaet Muenchen - Neurologische Klinik und Poliklinik, Munich
- Italy (3):
  - Universita' di Catania, Catania
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - University Hospital Friuli Centrale, Udine
- Great Ormond Street Hospital NHSFT, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No